CLINICAL TRIAL: NCT07304141
Title: Pharmacological Treatment - An Overview of Its Role in Managing Childhood Obesity
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Principal Investigator, Lovisa Sjogren, MD PhD, Göteborg University
Other Study IDs: Dnr 2023-04013-01
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Obesity (Disorder); Child Obesity
Keywords: liraglutide child obesity
MeSH Terms: conditions — Obesity; Pediatric Obesity | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study included adolescents aged 10-18 years with obesity who were offered liraglutide treatment
  Interventions: Other: Liraglutide 3 mg (Saxenda)

INTERVENTIONS:
Other: Liraglutide 3 mg (Saxenda) — This is a retrospective observational study of adolescents aged 10-18 years with obesity who were offered liraglutide treatment at the Pediatric Clinic in Region Halland and at the Regional Childhood Obesity Center, Queen Silvia's Children's Hospital, Sahlgrenska University Hospital.

SUMMARY:
The aim of the study is to examine the effects of pharmacological treatment for obesity on BMI trajectories and metabolic markers among patients in routine clinical care. A retrospective observational study. By collecting and analysing real-life data from the first children and adolescents in Sweden who have been offered pharmacological treatment for obesity, the results can contribute to a better understanding of how these treatments function in practice.

DETAILED DESCRIPTION:
Aim

The aim of this sub-study is to evaluate the impact of liraglutide treatment on the trajectory of body mass index (BMI), including BMI according to International Obesity Task Force (IOTF) criteria and BMI standard deviation score (BMI SDS), as well as its effects on cardiovascular risk markers among children and adolescents treated with liraglutide in two Swedish regions. The study seeks to generate real-world evidence on the effectiveness of liraglutide in routine clinical practice.

Study Design

This is a retrospective, observational study based on medical records of children and adolescents who received multidisciplinary obesity care for at least one year and were treated with liraglutide during 2022-2023 at either the Pediatric Clinic in Region Halland or the Regional Childhood Obesity Center at Queen Silvia's Children's Hospital. The study is non-interventional and does not introduce any additional risks beyond standard clinical care. Participation was voluntary, with informed consent obtained from legal guardians and assent from children.

Participants

Eligible participants include children and adolescents who:

Were enrolled in multidisciplinary obesity care for at least one year

Received liraglutide treatment during 2022-2023 at one of the study sites

Were invited to participate either during clinical visits or via written invitation

Data on comorbidities, including neuropsychiatric diagnoses, were also collected to assess potential confounding factors.

Data Collection

Data were extracted retrospectively from medical records and include:

Demographics: sex, age

Anthropometrics: height, weight, BMI, BMI SDS, BMI according to IOTF criteria

Treatment details: titration period, maximum tolerated dose, and treatment outcomes at 3-6, 12, 18.

Metabolic parameters: blood pressure, lipid profile, fasting glucose, and HbA1c

Comorbidities: neuropsychiatric and other relevant diagnoses

All data were anonymized and handled in accordance with Swedish data protection regulations.

Statistical Analysis

Descriptive Statistics:

Continuous variables (e.g., age, BMI, metabolic parameters) will be summarized using mean ± standard deviation (SD) or median with interquartile range (IQR), as appropriate.

Categorical variables (e.g., sex, comorbidities) will be summarized using counts and percentages.

Treatment effects at 3-6, 12, 18, and 24 months will be evaluated using appropriate repeated measures models, accounting for potential confounders such as age, sex, baseline BMI, and comorbidities.

Handling of Missing Data:

Missing data will be assessed for patterns and mechanisms.

Multiple imputation or sensitivity analyses may be performed depending on the proportion and nature of missing values.

Statistical Collaboration:

All analyses will be conducted in collaboration with an experienced statistician.

The analysis plan and results will be reviewed and validated by both the statistician and study supervisors.

Ethical Considerations

Participation was voluntary and did not affect ongoing clinical care.

Informed consent was obtained from legal guardians, with assent from children.

Data were anonymized and managed according to Swedish data protection laws.

The study was retrospective and non-interventional; no specific approval from the Swedish Medical Products Agency was required.

All procedures adhere to the ethical principles of the Declaration of Helsinki.

Dissemination

Results will be disseminated through a peer-reviewed publication and scientific conference presentations. Sub-study III is expected to be finalized in 2026.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 10-18 years with obesity who were offered pharmacological treatment
* Provided consent to participate
* Participants with short treatment duration, early adverse effects, or who proceeded to surgery are also included in baseline data

Exclusion Criteria:

* Hypothalamic obesity
* Craniopharyngioma
* Syndromic obesity / monogenic obesity

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children at the Pediatric Clinic, Region Halland, and at the Regional Childhood Obesity Center, Queen Silvia's Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Change in BMI SDS over time | The primary outcome, change in BMI SDS, will be evaluated at -12 months (pre-baseline), at baseline (0 months), and at +3-6, +12, and +18 months following treatment initiation.

CONTACTS AND LOCATIONS:
Locations (1):
- the Regional Childhood Obesity Center, Queen Silvia's Children's Hospital., Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers. This decision is based on ethical and legal considerations, as the dataset includes sensitive health information from children and adolescents. According to Swedish data protection regulations and the conditions of the ethical approval, IPD cannot be shared outside the research team. Only aggregated, anonymized results will be made available through scientific publications and presentations.